CLINICAL TRIAL: NCT04057677
Title: Exercise Training as an Intervention to Improve Muscle Function and Recovery Following Bed Rest in Older Adults With Type 2 Diabetes
Acronym: RECOVER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funds.
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1461891; R01AG060153 (NIH)
Record Dates: First submitted 2019-08-06; First posted 2019-08-15 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes; Muscular Atrophy; Sedentary Behavior; Exercise; Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Muscular Atrophy; Sedentary Behavior; Motor Activity; Glucose Intolerance | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The proposed clinical study is a prospective, parallel two arm, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Recovery (Experimental): Older males and females with pre-diabetes or type 2 diabetes. We are examining the effects of a recovery exercise program for older adults with pre-diabetes and type 2 diabetes. Following 10 days of bed rest and during the first 4 weeks of recovery, participants will perform a combination of aerobic and resistance exercise training.
  Interventions: Behavioral: Bed Rest Intervention; Behavioral: Exercise Program
- Non-Exercise Recovery (Experimental): Older males and females with pre-diabetes or type 2 diabetes. Participants in the ambulatory recovery group will not receive any exercise intervention or advice on exercise following 10 days of bed rest. Rather these participants will return to their regular daily routine that they engaged in prior to the bed rest intervention.
  Interventions: Behavioral: Bed Rest Intervention

INTERVENTIONS:
Behavioral: Bed Rest Intervention — The participant will remain in bed rest for 10 days at the clinical research unit at TRI, AdventHealth, Orlando.
Behavioral: Exercise Program — During the first 4 weeks following bed rest, participants will perform a combination of aerobic and resistance exercise training with a certified exercise physiologist 3 days per week at the TRI exercise training facility.
  Arms: Exercise Recovery

SUMMARY:
The purpose of this research is to gather data on how exercise can help recovery of muscle mass, strength, and physical function after bedrest in older adults with pre-diabetes and type 2 diabetes.

DETAILED DESCRIPTION:
Older adults with type 2 diabetes (T2D) experience an accelerated rate of sarcopenia, which is the deterioration in muscle mass, strength, and physical performance. Periods of disuse caused by illness or hospitalization causes rapid loss of muscle mass and strength, which negatively impact physical function upon re-ambulation. Without adequate rehabilitation, physical function does not fully recover in older adults following disuse, reducing the quality of life and loss of independence.

In this study, participants will enter a 10-day strictly controlled bed rest intervention at the Translational Research Institute (TRI) clinical research unit. Participants are randomized to either a progressive 4-week aerobic and resistance training recovery program at the exercise training or an ambulatory recovery group.

The overall objective of this project is to determine how an exercise intervention can aid in recovery of muscle mass, strength and physical function following bed rest in older adults with pre-diabetes and T2D.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be male or female, ages 60 through 80 years of age.
2. Participant has pre-diabetes or has been diagnosed with type 2 diabetes and taking 0-3 oral hypoglycemic agents, which include DPP-4 inhibitors, Sulfonylureas and/or Metformin therapy, and has an Hgb A1C < 8.0%.

   1. Participants on Insulin, injectable incretin mimetics, SGLT2 inhibitors, and Thiazolidinediones will be excluded.
   2. Pre-Diabetics are defined as having an HgbA1c of greater than or equal to 5.7% and less 6.5%, or a fasting glucose of greater than or equal to 100 mg/dl and less than 126 mg/dl or has a glucose of greater than or equal to 140 mg/dl and less than 200mg/dl at the 2 hour blood draw during OGTT
3. Participant must have renal function with an estimated glomerular filtration rate (eGFR) > 45 ml/min/1.73m2 determined at screening.
4. Participant's triglyceride level is < 350 mg/dl and LDL cholesterol is ≤ 150 mg/dl at screening.
5. Participant states willingness to follow protocol as described, the prescribed activity level and completing any forms needed throughout the study.
6. Participant has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study.

Exclusion Criteria:

1. Participant has type 1 Diabetes.
2. BMI > 40.0 kg/m2
3. Participant is actively pursuing weight loss and/or lifestyle changes.
4. Participant has a history of pressure ulcers.
5. Participant has a stated history of Deep Vein Thrombosis (DVT), pulmonary embolism, or a known hypercoagulable condition, or other clotting or bleeding disorders.
6. History of gastrointestinal or intracranial hemorrhage.
7. History of stroke or cerebrovascular accident.
8. Recent history of major trauma (within 3 months).
9. Thrombocytopenia (<100,000/microL) or hyperkalemia (K > 5.2) on screening laboratory assay. May repeat lab value per PI discretion.
10. Untreated or poorly controlled hypertension (SBP > 150, DBP > 95), or hypotension (SBP <100 DBP <60)
11. Participant has hypothyroidism (TSH less than or equal to (0.5mIU/L) or hyperthyroidism TSH greater than or equal to 10mIU/L.
12. Participant has current infection (requiring prescription antimicrobial or antiviral medication, or hospitalization), or corticosteroid treatment (with the exception of inhaled or topical steroids) in the last 3 months prior to screening visit.
13. Participant is currently taking anti-inflammatory medication or has had anti-inflammatory medication within 1 week prior to screening (including over the counter formulations; e.g. Aleve, Motrin, ibuprofen, naproxen, low dose asprin).
14. Participant has had surgery requiring > 2 days of hospitalization in the last 1 month prior to screening visit.
15. Participant has an active malignancy or autoimmune disease.
16. Participant has current significantly impaired liver function in the opinion of the study Medical Investigator (mild asymptomatic fatty liver is acceptable), or hepatic enzyme tests are ≥ 2.5 times normal limit.
17. Participant has a chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV, per self-report.
18. Participant is an amputee and/or has presence of partial or full artificial limb.
19. Participant has had a significant cardiovascular event (e.g. myocardial infarction, stroke) ≤ 6 months prior to screening visit; or stated history of congestive heart failure; or participant has evidence of cardiovascular disease assessed during the ECG at screening. In the event of a positive stress test, participants are referred to their primary care physician. If the electrocardiogram (ECG) is determined to be a false positive, participant may be allowed to participate in study after confirmatory records obtained.
20. Participant currently has uncontrolled severe diarrhea, nausea or vomiting.
21. Participant has an obstruction of the gastrointestinal tract, inflammatory bowel disease, short bowel syndrome or other forms of gastrointestinal disease such as stage III or above gastroesophageal reflux disease, gastroparesis, peptic ulcer disease, celiac disease, intestinal dysmotility, diverticulitis, ischemic colitis and bariatric surgery.
22. Participant cannot abstain from alcohol for the pre-bed rest and bed rest portion of the study. For the recovery portion of the study the participant must agree to consume no more than ~14gm of alcohol per day (equivalent to ~ 1 glass of wine (4-5 oz 12% ABV) or ~bottle of beer (12 oz 5% ABV) /day).
23. Participant cannot refrain from taking medications/dietary supplements/herbals or substances that could modulate glucose metabolism (other than oral hypoglycemic medications), or are considered anabolic, or reduce weight (fat mass), or that may interact with low-molecular weight heparin or induce hypo- or hyper-coagulable state, in the opinion of the PI or medical investigator, starting one week prior to Pre-bed rest phase and over the entire course of the study. These include progestational agents (except prescribed birth control), steroids, growth hormone, dronabinol, marijuana, calcium-beta-hydroxy-betamethylbutyrate (CaHMB), free amino acid supplements and dietary supplements to aid weight loss.
24. Participant has a mini-Mental State Examination score < 21.
25. Subjects who fulfill any of the contraindications for MRI; examples include metal implants, devices, paramagnetic objects contained within the body and excessive or metal-containing tattoos.
26. Unable to participate in MR or DEXA assessments due to physical limitations of equipment tolerances (e.g., MRI bore size and DEXA 450-pound weight limit), claustrophobia, or based on Investigator's judgment at screening.
27. Participant has a sensitivity or allergy to lidocaine.
28. Participant has a sensitivity or allergy to heparin, enoxaparin, or other low molecular weight heparin.
29. History of allergy to pork products.
30. History of heparin-induced thrombocytopenia.
31. Hemoglobin < 10.0 g/dL for females; < 11.0 g/dL for males; or participant has clinically significant signs/symptoms of anemia in the opinion of the PI or medical provider.
32. Concomitant medications with known contraindication or interaction with low-molecular weight heparin (including anti-platelet agents, anti-coagulant agents, non-steroidal anti-inflammatory drugs)
33. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete the study.
34. Participant experiences symptoms of claudication. Symptoms include cramping pain in the legs and/or difficulty walking.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Leg Lean Mass | Immediately following bed rest, and following the exercise or non-exercise recovery phase
  Determined by DXA (dual energy x-ray absorptiometry)
Mitochondrial Respiration | mmediately following bed rest, and following the exercise or non-exercise recovery phase
  Determined by high resolution respirometry in permeabilized muscle fiber bundles

SECONDARY OUTCOMES:
Insulin Sensitivity | mmediately following bed rest, and following the exercise or non-exercise recovery phase
  Determined by hyperinsulinemic euglycemic glucose clamp
Physical function | mmediately following bed rest, and following the exercise or non-exercise recovery phase
  Determined by short physical performance battery

CONTACTS AND LOCATIONS:
Overall Officials: Paul Coen, PhD, Principal Investigator — Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

REFERENCES:
- See also: AdventHealth Translational Research Institute — https://www.adventhealthresearchinstitute.com/research/translational-research-metabolism-diabetes

DOCUMENTS (1):
  • Study Protocol (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT04057677/Prot_001.pdf